CLINICAL TRIAL: NCT04773093
Title: Continous Intravenous Lidocaine Infusion Intraoperative for Craniotomy Tumor Removal Surgery: Effect to Brain Relaxation, Opioid Consumption and Postoperative Cognitive Status
Brief Title: Effect of Continous Intravenous Lidocaine Infusion Intraoperative for Craniotomy Tumor Removal Surgery
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, Susilo Chandra, MD, FRCA, Indonesia University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IndonesiaUAnes057
Record Dates: First submitted 2021-02-20; First posted 2021-02-26 (Actual); Last update posted 2021-02-26 (Actual); Status verified 2021-02

CONDITIONS: Craniotomy Tumor Removal Surgery
Keywords: intravenous lidocaine; craniotomy; brain relaxation; opioid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Continous Intravenous Lidocaine Infusion (Active Comparator): Patient will recieve Continous Intravenous Lidocaine Infusion
  Interventions: Drug: Continous Intravenous Lidocaine Infusion
- Placebo (Placebo Comparator): Patient will recieve placebo (NaCl 0.9% infusion)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Continous Intravenous Lidocaine Infusion — Patient will recieve intravenous Lidocaine dose 1.5 mg/kg at the time of induction and after that will receive maintenance by continous intravenous Lidocaine infusion dose 2 mg/kg/hour until the completion of surgery
  Arms: Continous Intravenous Lidocaine Infusion
Drug: Placebo — Patient will recieve Placebo NaCl 0.9% continuous intravenous infusion until the completion of surgery
  Arms: Placebo

SUMMARY:
This study aimed to compare continous intravenous lidocaine infusion and placebo on the effect to brain relaxation, opioid consumption and postoperative cognitive status in adult patient undergoing craniotomy tumor removal surgery

DETAILED DESCRIPTION:
Fifty subjects were given informed consent one day before surgery and then randomized into two groups: continous intravenous Lidocaine intraoperative and Placebo. Patient, the Anesthesist as data collector, and the Neurosurgeon as the outcome assessor are blinded to the randomization and the intervention given. Non invasive blood pressure, ECG, and pulse oxymetry monitor were set on the subject in the operating room. General anesthesia induction was done by Fentanyl 3 mcg/kg, Lidocaine 1.5 mg/kg or Placebo (according to allocation group), Propofol 1-2 mg/kg and Rocuronium 1 mg/kg. After the intubation, maintenance continous intravenous Lidocain dose 2 mg/kg/hours or Placebo were set until the completion of surgery. Other than intervention (Lidocain or Placebo), maintenance was done by volatile Sevoflurane 0.8 -1.0 MAC, intermittent Fentanyl, continous Atracurium dose 5 mcg/kg/minutes and Manitol 20% dose 0.5 g/kg 30 minutes before Neurosurgeon reach the duramater. At the time Neurosurgeon reach the duramater, before and after they open the duramater, Neurosurgeon will assess brain relaxation by direct inspection and palpation. Total Fentanyl intraoperative will record and Cognitive status pre and postoperative will assess using MMSE. Postoperatively patient will transport to the ICU for monitoring.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient age 18-65 years old undergo craniotomy tumor removal surgery
* Physical status ASA 1-3
* Compos mentis (GCS 15)
* Operation using pin head fixation

Exclusion Criteria:

* Patient or family refused to participate
* Has Atrioventricular block rhytm on ECG
* Has sign of circulation shock
* Midline shift > 5.4 mm on brain imaging
* Diagnose with Glioblastoma multiforme or Metastatic
* Vascular surgery
* Using CSF drainage (EVD, VP shunt, or Lumbal drain)
* Routine using or in treatmet using adrenergic agonist or antagonist drugs
* Routine consumption of opioid in last two weeks before surgery
* History of Local anesthetic hypersensitivity

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Brain relaxation | Up to 1 minute after duramater opening
  Measure by direct inspection and palpation of duramater and brain by Neurosurgeon. The result is using four points scale, grading the brain as completely relaxed, satisfactorily relaxed, firm and bulging
Preoperative cognitive status | During preanesthesia assessment
  Measured by using MMSE questionnaire
Postoperative cognitive status | 24-hours after surgery
  Measured by using MMSE questionnaire
Postoperative cognitive status | 36-hours after surgery
  Measured by using MMSE questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- National General Hospital Dr. Cipto Mangunkusumo, Jakarta Pusat, Indonesia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] de Robles P, Fiest KM, Frolkis AD, Pringsheim T, Atta C, St Germaine-Smith C, Day L, Lam D, Jette N. The worldwide incidence and prevalence of primary brain tumors: a systematic review and meta-analysis. Neuro Oncol. 2015 Jun;17(6):776-83. doi: 10.1093/neuonc/nou283. Epub 2014 Oct 13. PMID 25313193
- [Result] Fox BD, Cheung VJ, Patel AJ, Suki D, Rao G. Epidemiology of metastatic brain tumors. Neurosurg Clin N Am. 2011 Jan;22(1):1-6, v. doi: 10.1016/j.nec.2010.08.007. PMID 21109143
- [Result] Dunn LK, Durieux ME. Perioperative Use of Intravenous Lidocaine. Anesthesiology. 2017 Apr;126(4):729-737. doi: 10.1097/ALN.0000000000001527. No abstract available. PMID 28114177
- [Result] Weibel S, Jelting Y, Pace NL, Helf A, Eberhart LH, Hahnenkamp K, Hollmann MW, Poepping DM, Schnabel A, Kranke P. Continuous intravenous perioperative lidocaine infusion for postoperative pain and recovery in adults. Cochrane Database Syst Rev. 2018 Jun 4;6(6):CD009642. doi: 10.1002/14651858.CD009642.pub3. PMID 29864216
- [Result] Dunbar PJ, Visco E, Lam AM. Craniotomy procedures are associated with less analgesic requirements than other surgical procedures. Anesth Analg. 1999 Feb;88(2):335-40. doi: 10.1097/00000539-199902000-00021. PMID 9972752
- [Derived] Chandra S, Pryambodho P, Omega A. Evaluation of continuous intravenous lidocaine on brain relaxation, intraoperative opioid consumption, and surgeon's satisfaction in adult patients undergoing craniotomy tumor surgery: A randomized controlled trial. Medicine (Baltimore). 2022 Sep 9;101(36):e30216. doi: 10.1097/MD.0000000000030227. PMID 36086723